CLINICAL TRIAL: NCT03604393
Title: Increasing Human Papillomavirus (HPV) Immunization Rates: The Rural Adolescent Vaccine Enterprise (RAVE)
Brief Title: Increasing HPV Immunization Rates: The Rural Adolescent Vaccine Enterprise
Acronym: RAVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oregon Health and Science University (Other)
Collaborators: American Cancer Society, Inc. (Other); Oregon Health Authority (Other); University of Arkansas (Other)
Responsible Party: Principal Investigator, Lyle J. Fagnan, Director, Oregon Rural Practice-based Research Network (ORPRN), Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 18660
Record Dates: First submitted 2018-07-11; First posted 2018-07-27 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Human Papilloma Virus
Keywords: Immunization

STUDY DESIGN:
Intervention Model Description: Aims II and III are interventional, using a randomized stepped-wedge design with the practice as the unit of randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Practice Facilitation, Cluster 1 (Experimental): Intervention Cluster 1 is the first intervention arm designed to implement and test the effectiveness of a multi-component primary care practice-based intervention on initiation and completion of the HPV vaccine series as well as reduction in rates of missed opportunities to vaccinate.
  Interventions: Behavioral: Practice facilitation
- Practice Facilitation, Cluster 2 (Experimental): Intervention Cluster 2 is the second intervention arm designed to implement and test the effectiveness of a multi-component primary care practice-based intervention on initiation and completion of the HPV vaccine series as well as reduction in rates of missed opportunities to vaccinate.
  Interventions: Behavioral: Practice facilitation
- Practice Facilitation, Cluster 3 (Experimental): Intervention Cluster 3 is the third intervention arm designed to implement and test the effectiveness of a multi-component primary care practice-based intervention on initiation and completion of the HPV vaccine series as well as reduction in rates of missed opportunities to vaccinate.
  Interventions: Behavioral: Practice facilitation
- Practice Facilitation, Cluster 4 (Experimental): Intervention Cluster 4 is the fourth intervention arm designed to implement and test the effectiveness of a multi-component primary care practice-based intervention on initiation and completion of the HPV vaccine series as well as reduction in rates of missed opportunities to vaccinate.
  Interventions: Behavioral: Practice facilitation
- Practice Facilitation, Cluster 5 (Experimental): Intervention Cluster 5 is the final intervention arm designed to implement and test the effectiveness of a multi-component primary care practice-based intervention on initiation and completion of the HPV vaccine series as well as reduction in rates of missed opportunities to vaccinate.
  Interventions: Behavioral: Practice facilitation

INTERVENTIONS:
Behavioral: Practice facilitation — For this intervention, ORPRN Practice Facilitators will: 1) Build practice QI capacity by addressing the five Change Concepts; 2) Train practice clinicians and staff to generate reminder lists and notices in ALERT Immunization Information System (state immunization registry); 3) Develop an HPV immunization improvement plan for each practice using PDSA cycles and workflow mapping; and 4) Facilitate community engagement surrounding HPV vaccination messaging.

SUMMARY:
The goal of this study is to engage rural primary care clinics and community organizations to test interventions designed to increase HPV vaccinations in both male and female patients aged 9-26 years.

DETAILED DESCRIPTION:
The overarching goal of this study is to engage rural primary care clinics and community organizations to test interventions designed to increase HPV vaccinations in both male and female patients aged 9-26 years. Using a step-wedge randomized controlled trial, we will design and test the effectiveness of multi-component primary care practice-based interventions on the completion of the HPV vaccine series and will explore implementation timing in high and low functioning practices to determine how specific characteristics affect the delivery of the full series. Additionally, we will design and test the impact of a community organization-based intervention intended to educate the public about HPV and cancer risk and risk reduction via vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Oregon family medicine and pediatric clinics located in rural communities that see adequate numbers of patients in the age range we are studying (age 11-17 years).

Exclusion Criteria:

* We will not include neonates, decisionally impaired adults, and prisoners in this study.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22000 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
HPV vaccine series completion | 3 months
  A primary outcome variable is the receipt rate of the full series of HPV vaccine among males and females aged 11-17 years. Practices will be block randomized in five waves every six months. Outcomes will be measured every three months in all clusters at every period, so that each cluster provides data points in both the control and intervention conditions. Practices in each wave will be stratified based on designation of pediatric or family medicine clinic to balance pediatric/family medicine clinics at each wave. Outcome data collection will be collected from Oregon's ALERT Immunization System beginning in quarter four and up to 17, for 14 longitudinal data collection points per practice.

CONTACTS AND LOCATIONS:
Overall Officials: Lyle J Fagnan, MD, Principal Investigator — Oregon Health and Science University; Patty Carney, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- ORPRN, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Munoz N, Castellsague X, Berrington de Gonzalez A, Gissmann L. Chapter 1: HPV in the etiology of human cancer. Vaccine. 2006 Aug 31;24 Suppl 3:S3/1-10. doi: 10.1016/j.vaccine.2006.05.115. Epub 2006 Jun 23. PMID 16949995
- [Background] Lowy DR, Schiller JT. Reducing HPV-associated cancer globally. Cancer Prev Res (Phila). 2012 Jan;5(1):18-23. doi: 10.1158/1940-6207.CAPR-11-0542. PMID 22219162
- [Background] Koutsky L. The epidemiology behind the HPV vaccine discovery. Ann Epidemiol. 2009 Apr;19(4):239-44. doi: 10.1016/j.annepidem.2009.01.023. PMID 19344861
- [Background] Centers for Disease Control and Prevention (CDC). National and state vaccination coverage among adolescents aged 13-17 years--United States, 2011. MMWR Morb Mortal Wkly Rep. 2012 Aug 31;61(34):671-7. PMID 22932301
- [Background] Reagan-Steiner S, Yankey D, Jeyarajah J, Elam-Evans LD, Singleton JA, Curtis CR, MacNeil J, Markowitz LE, Stokley S. National, Regional, State, and Selected Local Area Vaccination Coverage Among Adolescents Aged 13-17 Years--United States, 2014. MMWR Morb Mortal Wkly Rep. 2015 Jul 31;64(29):784-92. doi: 10.15585/mmwr.mm6429a3. PMID 26225476
- [Background] Briss PA, Rodewald LE, Hinman AR, Shefer AM, Strikas RA, Bernier RR, Carande-Kulis VG, Yusuf HR, Ndiaye SM, Williams SM. Reviews of evidence regarding interventions to improve vaccination coverage in children, adolescents, and adults. The Task Force on Community Preventive Services. Am J Prev Med. 2000 Jan;18(1 Suppl):97-140. doi: 10.1016/s0749-3797(99)00118-x. PMID 10806982
- [Background] Oster NV, McPhillips-Tangum CA, Averhoff F, Howell K. Barriers to adolescent immunization: a survey of family physicians and pediatricians. J Am Board Fam Pract. 2005 Jan-Feb;18(1):13-9. doi: 10.3122/jabfm.18.1.13. PMID 15709059
- [Background] Recommendations regarding interventions to improve vaccination coverage in children, adolescents, and adults. Task Force on Community Preventive Services. Am J Prev Med. 2000 Jan;18(1 Suppl):92-6. No abstract available. PMID 10806981
- [Background] Niccolai LM, Hansen CE. Practice- and Community-Based Interventions to Increase Human Papillomavirus Vaccine Coverage: A Systematic Review. JAMA Pediatr. 2015 Jul;169(7):686-92. doi: 10.1001/jamapediatrics.2015.0310. PMID 26010507
- [Background] Smulian EA, Mitchell KR, Stokley S. Interventions to increase HPV vaccination coverage: A systematic review. Hum Vaccin Immunother. 2016 Jun 2;12(6):1566-88. doi: 10.1080/21645515.2015.1125055. Epub 2016 Feb 2. PMID 26838959
- [Background] Petrosky E, Bocchini JA Jr, Hariri S, Chesson H, Curtis CR, Saraiya M, Unger ER, Markowitz LE; Centers for Disease Control and Prevention (CDC). Use of 9-valent human papillomavirus (HPV) vaccine: updated HPV vaccination recommendations of the advisory committee on immunization practices. MMWR Morb Mortal Wkly Rep. 2015 Mar 27;64(11):300-4. PMID 25811679
- [Background] Meites E, Kempe A, Markowitz LE. Use of a 2-Dose Schedule for Human Papillomavirus Vaccination - Updated Recommendations of the Advisory Committee on Immunization Practices. MMWR Morb Mortal Wkly Rep. 2016 Dec 16;65(49):1405-1408. doi: 10.15585/mmwr.mm6549a5. PMID 27977643
- [Background] Jacobson RM, Rogacki B, Thompson DM, Roberts JR, Margolis B, Darden PM. Vaccination Rates among Adolescents in Minnesota as Compared with the United States: Not "Above Average". Minn Med. 2015 Nov-Dec;98(11-12):38-43. PMID 26720941
- [Background] Kepka D, Spigarelli MG, Warner EL, Yoneoka Y, McConnell N, Balch A. Statewide analysis of missed opportunities for human papillomavirus vaccination using vaccine registry data. Papillomavirus Res. 2016 Dec;2:128-132. doi: 10.1016/j.pvr.2016.06.002. PMID 27540595
- [Background] Roberts JR, Naifeh M, Jacobson RM, Hinton E, O'Brien E, Rogacki B, Thompson D, Margolis B, Darden PM. Adolescent Vaccination Performance in South Carolina Compared to the United States. J S C Med Assoc. 2015 Dec-2016 Jan;111(4):117-21. PMID 27141702
- [Background] Brewer NT, Fazekas KI. Predictors of HPV vaccine acceptability: a theory-informed, systematic review. Prev Med. 2007 Aug-Sep;45(2-3):107-14. doi: 10.1016/j.ypmed.2007.05.013. Epub 2007 Jun 2. PMID 17628649
- [Background] Marlow LA, Waller J, Wardle J. Parental attitudes to pre-pubertal HPV vaccination. Vaccine. 2007 Mar 1;25(11):1945-52. doi: 10.1016/j.vaccine.2007.01.059. Epub 2007 Jan 22. PMID 17284337
- [Background] Roberts JR, Thompson D, Rogacki B, Hale JJ, Jacobson RM, Opel DJ, Darden PM. Vaccine hesitancy among parents of adolescents and its association with vaccine uptake. Vaccine. 2015 Mar 30;33(14):1748-55. doi: 10.1016/j.vaccine.2015.01.068. Epub 2015 Feb 7. PMID 25659278
- [Background] Katz ML, Reiter PL, Heaner S, Ruffin MT, Post DM, Paskett ED. Acceptance of the HPV vaccine among women, parents, community leaders, and healthcare providers in Ohio Appalachia. Vaccine. 2009 Jun 19;27(30):3945-52. doi: 10.1016/j.vaccine.2009.04.040. Epub 2009 May 3. PMID 19389447
- [Background] Coyne CA, Demian-Popescu C, Friend D. Social and cultural factors influencing health in southern West Virginia: a qualitative study. Prev Chronic Dis. 2006 Oct;3(4):A124. Epub 2006 Sep 15. PMID 16978499
- [Background] Ferrer HB, Trotter C, Hickman M, Audrey S. Barriers and facilitators to HPV vaccination of young women in high-income countries: a qualitative systematic review and evidence synthesis. BMC Public Health. 2014 Jul 9;14:700. doi: 10.1186/1471-2458-14-700. PMID 25004868
- [Background] Lyttle NL, Stadelman K. Assessing awareness and knowledge of breast and cervical cancer among Appalachian women. Prev Chronic Dis. 2006 Oct;3(4):A125. Epub 2006 Sep 15. PMID 16978500
- [Background] Elnicki DM, Morris DK, Shockcor WT. Patient-perceived barriers to preventive health care among indigent, rural Appalachian patients. Arch Intern Med. 1995 Feb 27;155(4):421-4. PMID 7848026
- [Background] Thomas T, Blumling A, Delaney A. The Influence of Religiosity and Spirituality on Rural Parents' Health Decision Making and Human Papillomavirus Vaccine Choices. ANS Adv Nurs Sci. 2015 Oct-Dec;38(4):E1-E12. doi: 10.1097/ANS.0000000000000094. PMID 26517344
- [Background] Darden PM, Thompson DM, Roberts JR, Hale JJ, Pope C, Naifeh M, Jacobson RM. Reasons for not vaccinating adolescents: National Immunization Survey of Teens, 2008-2010. Pediatrics. 2013 Apr;131(4):645-51. doi: 10.1542/peds.2012-2384. Epub 2013 Mar 18. PMID 23509163
- [Background] Darden PM, Taylor JA, Brooks DA, Hendricks JW, Massoudi M, Stevenson JM, Bocian AB. How should immunization rates be measured in the office setting? A study from PROS and NMA PedsNet. Clin Pediatr (Phila). 2008 Apr;47(3):252-60. doi: 10.1177/0009922807308743. Epub 2007 Dec 5. PMID 18057163
- [Background] Slora EJ, Steffes JM, Harris D, Clegg HW, Norton D, Darden PM, Sullivan SA, Wasserman RC. Improving pediatric practice immunization rates through distance-based quality improvement: a feasibility trial from PROS. Clin Pediatr (Phila). 2008 Jan;47(1):25-36. doi: 10.1177/0009922807304597. Epub 2007 Aug 10. PMID 17693592
- [Background] McElligott JT, Darden PM. Are patient-held vaccination records associated with improved vaccination coverage rates? Pediatrics. 2010 Mar;125(3):e467-72. doi: 10.1542/peds.2009-0835. Epub 2010 Feb 15. PMID 20156897
- [Background] Mennito SH, Darden PM. Impact of practice policies on pediatric immunization rates. J Pediatr. 2010 Apr;156(4):618-22. doi: 10.1016/j.jpeds.2009.10.046. Epub 2010 Jan 13. PMID 20056238
- [Background] Darden PM, Gustafson KK, Nietert PJ, Jacobson RM. Extra-immunization as a clinical indicator for fragmentation of care. Public Health Rep. 2011 Jul-Aug;126 Suppl 2(Suppl 2):48-59. doi: 10.1177/00333549111260S207. PMID 21812169
- [Background] Fagnan LJ, Dorr DA, Davis M, McGinnis P, Mahler J, King MM, Michaels L. Turning on the care coordination switch in rural primary care: voices from the practices--clinician champions, clinician partners, administrators, and nurse care managers. J Ambul Care Manage. 2011 Jul-Sep;34(3):304-18. doi: 10.1097/JAC.0b013e31821c63ee. PMID 21673531
- [Background] Carney PA, Cook AJ, Miglioretti DL, Feig SA, Bowles EA, Geller BM, Kerlikowske K, Kettler M, Onega T, Elmore JG. Use of clinical history affects accuracy of interpretive performance of screening mammography. J Clin Epidemiol. 2012 Feb;65(2):219-30. doi: 10.1016/j.jclinepi.2011.06.010. Epub 2011 Oct 15. PMID 22000816
- [Background] Westfall JM, Mold J, Fagnan L. Practice-based research--"Blue Highways" on the NIH roadmap. JAMA. 2007 Jan 24;297(4):403-6. doi: 10.1001/jama.297.4.403. No abstract available. PMID 17244837
- [Background] Fagnan LJ, Morris C, Shipman SA, Holub J, King A, Angier H. Characterizing a practice-based research network: Oregon Rural Practice-Based Research Network (ORPRN) survey tools. J Am Board Fam Med. 2007 Mar-Apr;20(2):204-19. doi: 10.3122/jabfm.2007.02.060140. PMID 17341758
- [Background] Dietrich AJ, Carney PA, Winchell CW, Sox CH, Reed SC. An office systems approach to cancer prevention in primary care. Cancer Pract. 1997 Nov-Dec;5(6):375-81. PMID 9397706
- [Background] Dietrich AJ, Woodruff CB, Carney PA. Changing office routines to enhance preventive care. The preventive GAPS approach. Arch Fam Med. 1994 Feb;3(2):176-83. doi: 10.1001/archfami.3.2.176. PMID 7848489
- [Background] Dietrich AJ, O'Connor GT, Keller A, Carney PA, Levy D, Whaley FS. Cancer: improving early detection and prevention. A community practice randomised trial. BMJ. 1992 Mar 14;304(6828):687-91. doi: 10.1136/bmj.304.6828.687. PMID 1571644
- [Background] Carney PA, Dietrich AJ, Keller A, Landgraf J, O'Connor GT. Tools, teamwork, and tenacity: an office system for cancer prevention. J Fam Pract. 1992 Oct;35(4):388-94. PMID 1402726
- [Background] Cates JR, Diehl SJ, Crandell JL, Coyne-Beasley T. Intervention effects from a social marketing campaign to promote HPV vaccination in preteen boys. Vaccine. 2014 Jul 16;32(33):4171-8. doi: 10.1016/j.vaccine.2014.05.044. Epub 2014 Jun 2. PMID 24886960
- [Background] Cates JR, Shafer A, Diehl SJ, Deal AM. Evaluating a County-Sponsored Social Marketing Campaign to Increase Mothers' Initiation of HPV Vaccine for their Pre-teen Daughters in a Primarily Rural Area. Soc Mar Q. 2011 Spring;17(1):4-26. doi: 10.1080/15245004.2010.546943. PMID 21804767
- [Background] Moss JL, Gilkey MB, Rimer BK, Brewer NT. Disparities in collaborative patient-provider communication about human papillomavirus (HPV) vaccination. Hum Vaccin Immunother. 2016 Jun 2;12(6):1476-83. doi: 10.1080/21645515.2015.1128601. Epub 2016 Jan 19. PMID 26786888
- [Background] Keating KM, Brewer NT, Gottlieb SL, Liddon N, Ludema C, Smith JS. Potential barriers to HPV vaccine provision among medical practices in an area with high rates of cervical cancer. J Adolesc Health. 2008 Oct;43(4 Suppl):S61-7. doi: 10.1016/j.jadohealth.2008.06.015. PMID 18809147
- [Background] Hughes CC, Jones AL, Feemster KA, Fiks AG. HPV vaccine decision making in pediatric primary care: a semi-structured interview study. BMC Pediatr. 2011 Aug 30;11:74. doi: 10.1186/1471-2431-11-74. PMID 21878128
- [Background] Pope CA, Escobar-Gomez M, Davis BH, Roberts JR, O'Brien ES, Hinton E, Darden PM. The challenge of tetradic relationships in medically interpreted pediatric primary care visits: A descriptive study of communication practices. Patient Educ Couns. 2016 Apr;99(4):542-548. doi: 10.1016/j.pec.2015.10.032. Epub 2015 Dec 8. PMID 26796067
- [Background] Cabana MD, Rand CS, Powe NR, Wu AW, Wilson MH, Abboud PA, Rubin HR. Why don't physicians follow clinical practice guidelines? A framework for improvement. JAMA. 1999 Oct 20;282(15):1458-65. doi: 10.1001/jama.282.15.1458. PMID 10535437
- [Background] Stone EG, Morton SC, Hulscher ME, Maglione MA, Roth EA, Grimshaw JM, Mittman BS, Rubenstein LV, Rubenstein LZ, Shekelle PG. Interventions that increase use of adult immunization and cancer screening services: a meta-analysis. Ann Intern Med. 2002 May 7;136(9):641-51. doi: 10.7326/0003-4819-136-9-200205070-00006. PMID 11992299
- [Background] Dietrich AJ, Tobin JN, Cassells A, Robinson CM, Greene MA, Sox CH, Beach ML, DuHamel KN, Younge RG. Telephone care management to improve cancer screening among low-income women: a randomized, controlled trial. Ann Intern Med. 2006 Apr 18;144(8):563-71. doi: 10.7326/0003-4819-144-8-200604180-00006. PMID 16618953
- [Background] McPhee SJ, Detmer WM. Office-based interventions to improve delivery of cancer prevention services by primary care physicians. Cancer. 1993 Aug 1;72(3 Suppl):1100-12. doi: 10.1002/1097-0142(19930801)72:3+3.0.co;2-n. PMID 8334665
- [Background] Carney PA, O'Malley J, Buckley DI, Mori M, Lieberman DA, Fagnan LJ, Wallace J, Liu B, Morris C. Influence of health insurance coverage on breast, cervical, and colorectal cancer screening in rural primary care settings. Cancer. 2012 Dec 15;118(24):6217-25. doi: 10.1002/cncr.27635. Epub 2012 May 30. PMID 22648383
- [Background] Fagnan LJ, Shipman SA, Gaudino JA, Mahler J, Sussman AL, Holub J. To give or not to give: Approaches to early childhood immunization delivery in Oregon rural primary care practices. J Rural Health. 2011 Winter;27(4):385-93. doi: 10.1111/j.1748-0361.2010.00356.x. Epub 2011 Jan 11. PMID 21967382
- [Background] Solberg LI, Kottke TE, Brekke ML, Magnan S, Davidson G, Calomeni CA, Conn SA, Amundson GM, Nelson AF. Failure of a continuous quality improvement intervention to increase the delivery of preventive services. A randomized trial. Eff Clin Pract. 2000 May-Jun;3(3):105-15. PMID 11182958
- [Background] Miller WL, Crabtree BF, McDaniel R, Stange KC. Understanding change in primary care practice using complexity theory. J Fam Pract. 1998 May;46(5):369-76. PMID 9597994
- [Derived] Dickinson C, Bumatay S, Valenzuela S, Hatch BA, Carney PA. An Exploratory Study of Rural Parents' Knowledge and Attitudes About HPV Vaccination Following a Healthcare Visit With Their Child's Primary Care Provider. J Prim Care Community Health. 2023 Jan-Dec;14:21501319231201227. doi: 10.1177/21501319231201227. PMID 37933546
- [Derived] Carney PA, Hatch B, Stock I, Dickinson C, Davis M, Larsen R, Valenzuela S, Marino M, Darden PM, Gunn R, Ferrara L, Fagnan LJ. A stepped-wedge cluster randomized trial designed to improve completion of HPV vaccine series and reduce missed opportunities to vaccinate in rural primary care practices. Implement Sci. 2019 Mar 14;14(1):30. doi: 10.1186/s13012-019-0871-9. PMID 30866981

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-10): https://cdn.clinicaltrials.gov/large-docs/93/NCT03604393/Prot_SAP_000.pdf